CLINICAL TRIAL: NCT01039376
Title: A Phase III, Open Label, Randomized, Multicenter Trial of Ofatumumab Maintenance Treatment Versus no Further Treatment in Subjects With Relapsed Chronic Lymphocytic Leukemia (CLL) Who Have Responded to Induction Therapy
Brief Title: Ofatumumab Maintenance Treatment vs No Further Treatment in Relapsed CLL Responding to Induction Therapy
Acronym: PROLONG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 112517; COMB157C2301 (Other: Novartis)
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Results first posted 2015-04-21 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Leukaemia, Lymphocytic, Chronic
Keywords: maintenance therapy; anti-CD20 monoclonal antibody; ofatumumab
MeSH Terms: conditions — Leukemia, B-Cell | interventions — ofatumumab; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A: Ofatumumab (Experimental): 300 mg IV Week 1 followed by 1000 mg IV Week 2 1000 mg IV (a dose every 8 weeks for up to 2 years following the first 1000 mg dose)
  Interventions: Biological: Ofatumumab
- ARM B: Observation and assessments as per Arm A (Other): Disease status assessments to determine subject response or progression performed approximately every 8 weeks for up to 2 years for both arms according to IWCLL criteria
  Interventions: Other: Observation

INTERVENTIONS:
Biological: Ofatumumab — Ofatumumab for maintenance therapy as IV infusions every 8 weeks . The first dose was 300 mg followed 1 week later by 1000 mg and 1000 mg every 8 weeks thereafter for up to 2 years.
  Arms: ARM A: Ofatumumab
Other: Observation — Observation/Safety Evaluation
  Arms: ARM B: Observation and assessments as per Arm A

SUMMARY:
The purpose of this study was to determine if maintenance therapy with ofatumumab would prolong remission in patients with CLL who have responded to second or third line treatment. This study would also evaluate the safety of ofatumumab maintenance compared to observation (the current standard of care). This study was co-developed with the HOVON and NORDIC CLL group and would be conducted as a collaborative effort with GSK.

DETAILED DESCRIPTION:
The study met its primary objective at the protocol defined interim analysis (data cut-off 19-Jun-2014). The protocol-defined final analysis of the primary endpoint was performed when 280 PFS events were reached (data cut-off 20-Feb-2017).

ELIGIBILITY:
Inclusion Criteria:

* Adults with documented diagnosis of CLL based on the modified IWCLL updated NCI-WG guidelines (Hallek, 2008)
* At least PR according to the revised 2008 NCI-WG CLL criteria, within 3 months of the response assessment after the last dose of 2nd/3rd line treatment
* The anti-leukemic treatment before study entry should have been at least 3 months or 3 cycles
* ECOG Performance Status of 0-2
* Signed written informed consent prior to performing any study-specific procedures

Exclusion Criteria:

* Known primary or secondary fludarabine-refractory subjects, defined as treatment failure (failure to achieve a CR or PR) or disease progression within 6 months
* Prior maintenance therapy
* Known transformation of CLL (eg.Richter's transformation), prolymphocytic leukemia (PLL), or CNS involvement of CLL
* Active Autoimmune hemolytic anemia (AIHA) requiring treatment except if in the opinion of the investigator and medical monitor it is thought not to affect the subject's safety, the conduct of the study or the interpretation of the data
* Previous autologous or allogeneic stem cell transplantation
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis B or C
* Other past or current malignancy (with the exception of basal cell carcinoma or the skin or in situ carcinoma of the cervix or breasts) unless the tumor was successfully treated with curative intent at least 2 years prior to trial entry except if in the opinion of the investigator and medical monitor it is thought not to affect the subject's safety, the conduct of the study or the interpretation of the data
* Clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months prior to screening, congestive heart failure, and arrhythmia requiring therapy, with the exception of exta systoles or minor conduction abnormalities except if in the opinion of the investigator and medical monitor it is thought not to affect the subject's safety, the conduct of the study or the interpretation of the data
* History of significant cerebrovascular disease or event with symptoms or sequelae
* Significant concurrent, uncontrolled medical condition that in the opinion of the investigator or GSK medical monitor contraindicates participation in this study
* Other anti-leukemic use of medications including glucocorticoids
* Known HIV positive
* Screening laboratory values: platelets <50 x 10x9/L, neutrophils<1.0 x 10x9/L, Creatinine > 1.5 X upper normal limit (unless normal creatinine clearance), total bilirubin >1.5 X upper normal limit, ALT >2.5 X upper normal limit (unless due to liver involvement of CLL), alkaline phosphase > 2.5 X upper normal limit
* Known or suspected hypersensitivity to ofatumumab that in the opinion of the investigator or medical monitor contraindicates study participation
* Subjects who have received treatment with any non-marketed drug substance or experimental therapy within 5-terminal half-lives or 4 weeks whichever is longer prior to first dose of study medication or currently participating in any other interventional clinical study
* Lactating women, women with a positive pregnancy test at Visit 1 or women (of childbearing potential) as well as men with partners of childbearing potential, who are not willing to use adequate contraception from study start through one year following last ofatumumab dose. Adequate contraception is defined as abstinence, oral hormonal birth control, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, intrauterine device, and male partner sterilization if male partner is sole partner for that subject. For females in the USA, the use of a double barrier method is also considered adequate (condom or occlusive cap plus spermicidal agent).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2010-05-06 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (176):
- United States (40):
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Jonesboro, Arkansas
  - Novartis Investigative Site, Berkeley, California
  - Novartis Investigative Site, La Verne, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Pablo, California
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Lake Worth, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Pembroke Pines, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Post Falls, Idaho
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Westwood, Kansas
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Cumberland, Maryland
  - Novartis Investigative Site, Hagerstown, Maryland
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Chattanooga, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Orem, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
- Argentina (6):
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Derqui, Pilar, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
- Australia (5):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (7):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Wilrijk
- Brazil (5):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Goiania - GO, Goiás
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (6):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Czechia (5):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Pelhřimov
  - Novartis Investigative Site, Prague
- Denmark (3):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Roskilde
- Finland (5):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Pori
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (12):
  - Novartis Investigative Site, Blois
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Saint-Pierre
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Piraeus
  - Novartis Investigative Site, Thessaloniki
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Szeged
- India (3):
  - Novartis Investigative Site, Ahmedabad
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, Pune
- Israel (10):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Zrifin
- Italy (6):
  - Novartis Investigative Site, Modena, Emilia-Romagna
  - Novartis Investigative Site, Piacenza, Emilia-Romagna
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Novara, Piedmont
  - Novartis Investigative Site, Turin, Piedmont
  - Novartis Investigative Site, Pisa, Tuscany
- Netherlands (16):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Blaricum
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Dordrecht
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Hoofddorp
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Sittard-geleen
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Tilburg
- Novartis Investigative Site, Oslo, Norway
- Poland (6):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Słupsk
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, San Juan, Puerto Rico
- Russia (7):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, St'Petersburg
  - Novartis Investigative Site, Volgograd
- Novartis Investigative Site, Seoul, South Korea
- Spain (6):
  - Novartis Investigative Site, Hospitalet de Llobregat (Barcelona)
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Toledo
  - Novartis Investigative Site, Zaragoza
- Sweden (6):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- Ukraine (9):
  - Novartis Investigative Site, Cherkasy
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Khmelnytskyi
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Makiivka
  - Novartis Investigative Site, Vinnitsa
  - Novartis Investigative Site, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were stratified based on complete or partial remission at study entry, number of previous induction treatments (2 versus 3) and type of prior treatment (chemoimmunotherapy, only alkylating monotherapy, or other treatment). Participants were then randomized in a 1:1 ratio to receive ofatumumab or no further treatment.
Groups:
- Ofatumumab: Participants with relapsed CLL received IV infusions of ofatumumab on Day 1 (300 mg) and Day 8 (1000 mg) in the first cycle, followed by infusions of 1000 mg every 2 months for up to 2 years following the first 1000 mg dose.
- Observation: Participants with relapsed CLL received no treatment and were under observation for up to 2 years.
Period: Overall Study
Arm/Group | Ofatumumab | Observation
Started | 240 | 240
Completed | 110 | 114
Not Completed | 130 | 126
Not completed — Lost to Follow-up | 5 | 12
Not completed — Physician Decision | 15 | 10
Not completed — Withdrawal by Subject | 20 | 32
Not completed — Study terminated by Sponsor | 90 | 72

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included subjects who were randomized in the study. Subjects were grouped based on how they were randomized regardless of which treatment they received. This population was used for evaluation of all efficacy assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofatumumab | Observation | Total
Number analyzed (Participants) | 240 | 240 | 480
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 121 | 120 | 241
  >=65 years | 119 | 120 | 239
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (10.31) | 64.1 (9.61) | 64.0 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 80 | 159
  Male | 161 | 160 | 321
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 15 | 18 | 33
  Not Hispanic/Latino | 225 | 221 | 446
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival, as Assessed by the Investigator
Description: Progression-free survival is defined as the time from randomization to the date of disease progression (PD) or death due to any cause. PD was determined by the investigator according to the definitions of response in the International Workshop for Chronic Lymphocytic Leukemia (IWCLL) updated National Cancer Institute-Sponsored Working Group (NCI-WG) guidelines. According to the guidelines, PD is characterized by at least one of the following: lymphadenopathy (appearance of any new lesion such as enlarged lymph nodes (>1.5 centimeter [cm]), spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site); an increase by 50% or more in the previously noted enlargement of the liver or spleen; an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter; transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukemia.
Time Frame: From randomization until progression or death (up to 79 months)
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 240 | 240
Months | 34.17 [29.70 to 38.01] | 16.89 [12.98 to 20.37]
Statistical Analysis 1: Comparison: Ofatumumab vs Observation; Test type: Superiority; p < 0.0001, Stratified log rank test; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.43 to 0.70] — Hazard ratios were obtained using the Pike estimator. A hazard ratio of <1 indicated a lower risk with ofatumumab maintenance compared with no further treatment

2. Primary Outcome: Progression-free Survival, as Assessed by the Independent Review Committee (IRC)
Description: Progression-free survival is defined as the time from randomization to the date of disease progression (PD) or death due to any cause. PD was determined by the IRC according to the definitions of response in the International Workshop for Chronic Lymphocytic Leukemia (IWCLL) updated National Cancer Institute-Sponsored Working Group (NCI-WG) guidelines. According to the guidelines, PD is characterized by at least one of the following: lymphadenopathy (appearance of any new lesion such as enlarged lymph nodes (>1.5 centimeter [cm]), spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site); an increase by 50% or more in the previously noted enlargement of the liver or spleen; an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter; transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukemia.
Time Frame: From randomization until progression or death (up to 79 months)
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 240 | 240
Months | 33.74 [28.35 to 38.01] | 14.98 [11.63 to 19.12]
Statistical Analysis 1: Comparison: Ofatumumab vs Observation; Test type: Superiority; p < 0.0001, Stratified log rank test; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.42 to 0.68] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from randomization to date of death.
Time Frame: From randomization until death (up to 88 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 240 | 240
Months | NA [68.96 to NA] — There were not enough events on the survival curve to estimate a median or the upper limits of the confidence intervals. | 73.63 [66.53 to NA] — There were not enough events on the survival curve to estimate a median or the upper limits of the confidence intervals.
Statistical Analysis 1: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.6046, Stratified log rank test; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.69 to 1.25] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Improvement in Response From Baseline
Description: Improvement in response was assessed by calculating the percentage of participants who changed from partial response (PR) at Baseline to complete response during the study.
Time Frame: From Baseline until the end of the study (up to 88 months)
Population: ITT Population. Only participants who had PR at study entry were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 193 | 192
Participants | 16 | 8

5. Secondary Outcome: Time to Next Therapy
Description: Time to next therapy is defined as the time from randomization to the date of receiving the next CLL treatment.
Time Frame: From randomization until the end of the study (up to 88 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 240 | 240
Months | 36.21 [30.49 to 41.40] | 27.56 [23.49 to 32.49]
Statistical Analysis 1: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0178, Stratified log rank test; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.62 to 0.96] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Progression-free Survival After Next-line Therapy
Description: Progression-free survival after next-line therapy is defined as the time from randomization until progression or death following the next-line therapy and counted as events deaths prior to next-line therapy. Participants who received next-line therapy and who did not have progression or death after next-line therapy were censored at their last date of contact. Participant who died prior to next-line therapy, was counted as an event.
Time Frame: From randomization until progression or death (up to 88 months)
Population: ITT Population. Only participants who received next-line therapy and subjects who died prior to receiving next-line therapy were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 168 | 180
Months | NA [NA to NA] — There were not enough events for this endpoint to reach a median or confidence interval. | NA [NA to NA] — There were not enough events for this endpoint to reach a median or confidence interval.
Statistical Analysis 1: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.3136, log rank test; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.42 to 1.32] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time to Progression After Next-line Therapy
Description: Time to progression after next-line therapy is defined as the time from progression following randomization until progression or death following next-line therapy and counted as events deaths prior to next-line therapy. Participants who received next-line therapy with a PD prior to receiving next line therapy and who did not had progression or death after next-line therapy were censored at their last date of contact. If a participant died prior to next-line therapy, this was counted as an event.
Time Frame: From randomization until progression or death (up to 88 months)
Population: ITT Population. Only participants who received next-line therapy and who also had PD prior to next line therapy were analysed. Participants who died prior to next-line therapy were also included for analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 151 | 170
Months | NA [NA to NA] — There are not enough events for this endpoint to reach a median or confidence interval. | NA [NA to NA] — There are not enough events for this endpoint to reach a median or confidence interval.
Statistical Analysis 1: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.1603, log rank test; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.29 to 1.19] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline (BL) in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Chronic Lymphocytic Leukaemia 16 Item Module (EORTC QLQ-CLL 16)
Description: The EORTC QLQ-CLL16 is comprised of 16 questions that address 5 domains of health-related quality of life (HRQoL) important in CLL. There are 4 multi-item scales - fatigue (2 items), treatment side effects ([TSE], 4 items), disease symptoms (disease effects scale [DES], 4 items), and infection (4 items) - and single-item scales (social activities [Social Problems (SP) Scale] and future health worries [Future Health (FH) Scale]). These are measured on a four-point Likert scale, where 1 = not at all and 4 = very much. These scores are transformed to give a rating from 0 - 100, where 0 = no symptoms or problems and 100 = severe symptoms or problems. Changes from Baseline were analyzed by a mixed model-repeated measures analysis of covariance (ANCOVA).
Time Frame: From randomization until the end of the study (up to 47 months)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 238 | 236
Scores on a scale
  Disease Effects Scale | 0.36 (1.81) | 2.56 (1.78)
  Fatigue Scale | -0.16 (2.96) | 3.63 (2.93)
  Future Health Scale | -8.66 (3.69) | -5.08 (3.65)
  Infection Scale | 0.77 (2.20) | 0.25 (2.17)
  Social Problems Scale | 5.69 (3.20) | 10.02 (3.16)
  Treatment Side Effects Scale | -0.54 (1.77) | 1.95 (1.74)
Statistical Analysis 1: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0199, Repeated measures analysis of covariance — The analysis is adjusted for BL score, actual strata, age group, BL ECOG performance status and Binet stage at Screening using mixed-model (Proc Mixed) repeated with intercept, BL score by time and treatment by time interaction; Mean Difference (Final Values) = -2.19, 95% CI 2-sided [-4.04 to -0.35] — Disease Effects Scale
Statistical Analysis 2: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0085, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -3.79, 95% CI 2-sided [-6.61 to -0.97] — Fatigue Scale
Statistical Analysis 3: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0642, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -3.58, 95% CI 2-sided [-7.37 to 0.21] — Future Health Scale
Statistical Analysis 4: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.6398, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-1.67 to 2.72] — Infection Scale
Statistical Analysis 5: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0055, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -4.32, 95% CI 2-sided [-7.37 to -1.28] — Social Problems Scale
Statistical Analysis 6: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0063, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -2.49, 95% CI 2-sided [-4.27 to -0.71] — Side Effects Scale

9. Secondary Outcome: Change From Baseline in the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Score
Description: The EORTC QLQ-C30 is a self-reported, 30-item cancer-specific instrument that assesses 15 domains: physical functioning (5 items), role functioning (2 items), emotional functioning (4 items), cognitive functioning (2 items), social functioning (2 items), pain (2 items), fatigue (3 items), nausea and vomiting (2 items), five single-item symptom scores (insomnia, loss of appetite, constipation, diarrhea, and dyspnea), a single item asking about financial difficulties, and global health status/quality of life (QOF) consisting of 2 items. Functional and symptoms scales were measured on a four-point Likert scale, where 1 = not at all and 4 = very much, whereas global health status or QOF was assessed using a 7-item Likert scale, ranging from "poor" (worse quality of life) to "excellent" (better quality of life). Changes from Baseline were analyzed by mixed model-repeated measures ANCOVA.
Time Frame: From randomization until the end of the study (up to 47 months)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 238 | 236
Scores on a scale
  Appetite Loss | -0.63 (2.33) | 0.85 (2.30)
  Cognitive Functioning | -1.63 (2.30) | -3.03 (2.29)
  Constipation | -1.71 (2.30) | 0.27 (2.27)
  Diarrhoea | -1.99 (2.23) | -2.49 (2.20)
  Dyspnoea | 0.44 (2.71) | 2.76 (2.67)
  Emotional Functioning | -0.83 (2.47) | -4.72 (2.44)
  Fatigue | -0.02 (2.89) | 4.61 (2.85)
  Financial Difficulties | 4.09 (3.31) | 5.85 (3.26)
  Nausea and Vomiting | 0.28 (1.12) | 1.50 (1.11)
  Pain | 1.82 (2.89) | 4.87 (2.87)
  Physical Functioning | -2.25 (2.01) | -4.07 (2.01)
  Global Health Status/QOL | -0.17 (2.52) | -1.94 (2.49)
  Role Functioning | -6.94 (3.04) | -10.51 (3.00)
  Social Functioning | -4.15 (2.71) | -7.80 (2.69)
  Insomnia | -4.49 (3.51) | -2.70 (3.48)
Statistical Analysis 1: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.1816, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.48, 95% CI 2-sided [-3.64 to 0.69] — Appetite Loss
Statistical Analysis 2: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.2863, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 1.40, 95% CI 2-sided [-1.18 to 3.97] — Cognitive Functioning
Statistical Analysis 3: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0932, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.97, 95% CI 2-sided [-4.28 to 0.33] — Constipation
Statistical Analysis 4: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.6533, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-1.67 to 2.66] — Diarrhoea
Statistical Analysis 5: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0963, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -2.32, 95% CI 2-sided [-5.06 to 0.42] — Dyspnoea
Statistical Analysis 6: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0037, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 3.89, 95% CI 2-sided [1.27 to 6.51] — Emotional Functioning
Statistical Analysis 7: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0013, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -4.63, 95% CI 2-sided [-7.45 to -1.82] — Fatigue
Statistical Analysis 8: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.2902, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-5.02 to 1.51] — Financial Difficulties
Statistical Analysis 9: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0606, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-2.49 to 0.05] — Nausea and Vomiting
Statistical Analysis 10: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0393, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -3.04, 95% CI 2-sided [-5.93 to -0.15] — Pain
Statistical Analysis 11: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0968, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 1.81, 95% CI 2-sided [-0.33 to 3.96] — Physical Functioning
Statistical Analysis 12: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.1449, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 1.78, 95% CI 2-sided [-0.61 to 4.17] — Global Health Status/QOL
Statistical Analysis 13: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0259, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 3.56, 95% CI 2-sided [0.43 to 6.70] — Role Functioning
Statistical Analysis 14: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0175, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 3.65, 95% CI 2-sided [0.64 to 6.65] — Social Functioning
Statistical Analysis 15: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.3209, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -1.79, 95% CI 2-sided [-5.33 to 1.75] — Insomnia

10. Secondary Outcome: Change From Baseline in the Quality of Life Status as Assessed by the EuroQol-5D (EQ-5D) Scale
Description: EQ-5D is comprised of a 5-item health status measure and a visual analogue scale (VAS) and is used to generate two scores: the utility score and the thermometer score. The utility score measures mobility, self-care, usual activities, pain, discomfort, and anxiety/depression. Responses to each of the 5 health states are measured on a 3-point scale (level 1 = no problem; level 2 = some or moderate problem[s] and level 3 = unable, or extreme problems). Responses are typically converted into health utilities or valuations on a scale ranging from 0 (worst health) to 1 (perfect health). The thermometer score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Changes from Baseline were analyzed by mixed model-repeated measures ANCOVA. A negative adjusted mean change from Baseline represents a worsening of quality of life.
Time Frame: From screening until the end of the study (up to 47 months)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 238 | 236
Scores on a scale
  Utility Score | -0.02 (0.03) | -0.05 (0.03)
  Thermometer Score | -0.37 (2.05) | -1.75 (2.04)
Statistical Analysis 1: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.0110, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [0.01 to 0.06] — Utility Score
Statistical Analysis 2: Comparison: Ofatumumab vs Observation; Test type: Superiority; p = 0.1999, Repeated measures analysis of covariance — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [-0.73 to 3.49] — Thermometer Score

11. Secondary Outcome: Number of Participants With an Improvement in Eastern Cooperative Oncology Group (ECOG) Performance Status at the Indicated Time Points
Description: Improvement is defined as a decrease from Baseline by at least one step on the ECOG performance status scale (improvement categorized as yes or no). Improvement in ECOG performance status was measured.
Time Frame: From randomization until the end of the study (up to 88 months)
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 240 | 240
Participants
  C1 W2/M1: number analyzed (Participants) | 234 | 202
  C1 W2/M1 | 10 | 12
  C2 W9/M3: number analyzed (Participants) | 226 | 222
  C2 W9/M3 | 20 | 17
  C3 W17/M5: number analyzed (Participants) | 214 | 203
  C3 W17/M5 | 16 | 17
  C4 W25/M7: number analyzed (Participants) | 200 | 184
  C4 W25/M7 | 18 | 16
  C5 W33/M9: number analyzed (Participants) | 194 | 171
  C5 W33/M9 | 16 | 18
  C6 W41/M11: number analyzed (Participants) | 183 | 151
  C6 W41/M11 | 14 | 12
  C7 W49/M13: number analyzed (Participants) | 174 | 137
  C7 W49/M13 | 18 | 14
  C8 W57/M15: number analyzed (Participants) | 154 | 119
  C8 W57/M15 | 14 | 15
  C9 W65/M17: number analyzed (Participants) | 140 | 107
  C9 W65/M17 | 11 | 12
  C10 W73/M19: number analyzed (Participants) | 136 | 103
  C10 W73/M19 | 14 | 10
  C11 W81/M21: number analyzed (Participants) | 124 | 94
  C11 W81/M21 | 10 | 9
  C12 W89/M23: number analyzed (Participants) | 119 | 82
  C12 W89/M23 | 11 | 7
  C13 W97/M25: number analyzed (Participants) | 112 | 79
  C13 W97/M25 | 9 | 7
  3M FU: number analyzed (Participants) | 106 | 63
  3M FU | 11 | 6
  6M FU: number analyzed (Participants) | 104 | 61
  6M FU | 9 | 4
  9M FU: number analyzed (Participants) | 92 | 50
  9M FU | 5 | 5
  12M FU: number analyzed (Participants) | 81 | 43
  12M FU | 6 | 5
  15M FU: number analyzed (Participants) | 66 | 39
  15M FU | 4 | 4
  18M FU: number analyzed (Participants) | 60 | 35
  18M FU | 4 | 3
  21M FU: number analyzed (Participants) | 51 | 32
  21M FU | 3 | 3
  24M FU: number analyzed (Participants) | 48 | 26
  24M FU | 3 | 2
  27M FU: number analyzed (Participants) | 40 | 24
  27M FU | 3 | 1
  30M FU: number analyzed (Participants) | 35 | 18
  30M FU | 3 | 1
  33M FU: number analyzed (Participants) | 30 | 17
  33M FU | 3 | 1
  36M FU: number analyzed (Participants) | 27 | 15
  36M FU | 3 | 1
  39M FU: number analyzed (Participants) | 22 | 12
  39M FU | 1 | 2
  42M FU: number analyzed (Participants) | 17 | 10
  42M FU | 0 | 0
  45M FU: number analyzed (Participants) | 14 | 7
  45M FU | 0 | 1
  48M FU: number analyzed (Participants) | 10 | 5
  48M FU | 0 | 1
  51M FU: number analyzed (Participants) | 8 | 4
  51M FU | 0 | 1
  54M FU: number analyzed (Participants) | 6 | 2
  54M FU | 1 | 1
  57M FU: number analyzed (Participants) | 3 | 2
  57M FU | 0 | 1
  60M FU: number analyzed (Participants) | 2 | 2
  60M FU | 0 | 1
  Withdrawal: number analyzed (Participants) | 79 | 94
  Withdrawal | 5 | 10
  Worst-Case Post Baseline: number analyzed (Participants) | 238 | 235
  Worst-Case Post Baseline | 3 | 5

12. Secondary Outcome: Number of Participants With the Indicated Constitutional or B-symptoms at the Indicated Time Points
Description: Participants with the indicated constitutional or B-symptoms (night sweats [without signs of infection]; unintentional weight loss >= 10% within the previous 6 months; recurrent, unexplained fever of > 38 degrees celcius or 100.5 degrees fahrenheit for 2 weeks; and extreme fatigue) were presented. The proportion of participants with no night sweats, no weight loss, no fever and no extreme fatigue were summarized.
Time Frame: From Screening until the end of the study (up to 88 months)
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT population.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 240 | 240
Participants
  SCR, extreme fatigue | 0 | 7
  SCR, fever | 0 | 1
  SCR, night sweats | 13 | 8
  SCR, weight loss | 2 | 1
  C1 W2/M1, extreme fatigue: number analyzed (Participants) | 236 | 204
  C1 W2/M1, extreme fatigue | 0 | 2
  C1 W2/M1, fever: number analyzed (Participants) | 236 | 204
  C1 W2/M1, fever | 0 | 0
  C1 W2/M1, night sweats: number analyzed (Participants) | 236 | 204
  C1 W2/M1, night sweats | 9 | 6
  C1 W2/M1, weight loss: number analyzed (Participants) | 236 | 204
  C1 W2/M1, weight loss | 4 | 1
  C2 W9/M3, extreme fatigue: number analyzed (Participants) | 227 | 223
  C2 W9/M3, extreme fatigue | 3 | 3
  C2 W9/M3, fever: number analyzed (Participants) | 227 | 223
  C2 W9/M3, fever | 1 | 2
  C2 W9/M3, night sweats: number analyzed (Participants) | 227 | 223
  C2 W9/M3, night sweats | 6 | 10
  C2 W9/M3, weight loss: number analyzed (Participants) | 227 | 223
  C2 W9/M3, weight loss | 3 | 1
  C3 W17/M5, extreme fatigue: number analyzed (Participants) | 215 | 206
  C3 W17/M5, extreme fatigue | 4 | 5
  C3 W17/M5, fever: number analyzed (Participants) | 215 | 206
  C3 W17/M5, fever | 1 | 2
  C3 W17/M5, night sweats: number analyzed (Participants) | 215 | 206
  C3 W17/M5, night sweats | 6 | 10
  C3 W17/M5, weight loss: number analyzed (Participants) | 215 | 206
  C3 W17/M5, weight loss | 3 | 3
  C4 W25/M7, extreme fatigue (n=203, 187): number analyzed (Participants) | 203 | 187
  C4 W25/M7, extreme fatigue (n=203, 187) | 1 | 3
  C4 W25/M7, fever: number analyzed (Participants) | 203 | 187
  C4 W25/M7, fever | 1 | 2
  C4 W25/M7, night sweats: number analyzed (Participants) | 203 | 187
  C4 W25/M7, night sweats | 5 | 7
  C4 W25/M7, weight loss: number analyzed (Participants) | 203 | 187
  C4 W25/M7, weight loss | 1 | 1
  C5 W33/M9, extreme fatigue: number analyzed (Participants) | 196 | 171
  C5 W33/M9, extreme fatigue | 1 | 5
  C5 W33/M9, fever: number analyzed (Participants) | 196 | 171
  C5 W33/M9, fever | 1 | 0
  C5 W33/M9, night sweats fatigue: number analyzed (Participants) | 196 | 171
  C5 W33/M9, night sweats fatigue | 7 | 8
  C5 W33/M9, weight loss: number analyzed (Participants) | 196 | 171
  C5 W33/M9, weight loss | 0 | 4
  C6 W41/M11, extreme fatigue: number analyzed (Participants) | 184 | 152
  C6 W41/M11, extreme fatigue | 1 | 2
  C6 W41/M11, fever: number analyzed (Participants) | 184 | 152
  C6 W41/M11, fever | 2 | 0
  C6 W41/M11, night sweats: number analyzed (Participants) | 184 | 152
  C6 W41/M11, night sweats | 7 | 7
  C6 W41/M11, weight loss: number analyzed (Participants) | 184 | 152
  C6 W41/M11, weight loss | 0 | 0
  C7 W49/M13, extreme fatigue: number analyzed (Participants) | 175 | 138
  C7 W49/M13, extreme fatigue | 1 | 1
  C7 W49/M13, fever: number analyzed (Participants) | 175 | 138
  C7 W49/M13, fever | 0 | 0
  C7 W49/M13, night sweats: number analyzed (Participants) | 175 | 138
  C7 W49/M13, night sweats | 3 | 5
  C7 W49/M13, weight loss: number analyzed (Participants) | 175 | 138
  C7 W49/M13, weight loss | 2 | 1
  C8 W57/M15, extreme fatigue: number analyzed (Participants) | 155 | 122
  C8 W57/M15, extreme fatigue | 1 | 1
  C8 W57/M15, fever: number analyzed (Participants) | 155 | 122
  C8 W57/M15, fever | 2 | 0
  C8 W57/M15, night sweats: number analyzed (Participants) | 155 | 122
  C8 W57/M15, night sweats | 4 | 4
  C8 W57/M15, weight loss: number analyzed (Participants) | 155 | 122
  C8 W57/M15, weight loss | 2 | 3
  C9 W65/M17, extreme fatigue: number analyzed (Participants) | 142 | 107
  C9 W65/M17, extreme fatigue | 2 | 2
  C9 W65/M17, fever: number analyzed (Participants) | 142 | 107
  C9 W65/M17, fever | 2 | 0
  C9 W65/M17, night sweats: number analyzed (Participants) | 142 | 107
  C9 W65/M17, night sweats | 7 | 4
  C9 W65/M17, weight loss: number analyzed (Participants) | 142 | 107
  C9 W65/M17, weight loss | 1 | 2
  C10 W73/M19, extreme fatigue: number analyzed (Participants) | 137 | 103
  C10 W73/M19, extreme fatigue | 2 | 2
  C10 W73/M19, fever: number analyzed (Participants) | 137 | 103
  C10 W73/M19, fever | 1 | 0
  C10 W73/M19, night sweats: number analyzed (Participants) | 137 | 103
  C10 W73/M19, night sweats | 7 | 4
  C10 W73/M19, weight loss: number analyzed (Participants) | 137 | 103
  C10 W73/M19, weight loss | 2 | 1
  C11 W81/M21, extreme fatigue: number analyzed (Participants) | 126 | 96
  C11 W81/M21, extreme fatigue | 0 | 3
  C11 W81/M21, fever: number analyzed (Participants) | 126 | 96
  C11 W81/M21, fever | 1 | 0
  C11 W81/M21, night sweats: number analyzed (Participants) | 126 | 96
  C11 W81/M21, night sweats | 2 | 4
  C11 W81/M21, weight loss: number analyzed (Participants) | 126 | 96
  C11 W81/M21, weight loss | 0 | 0
  C12 W89/M23, extreme fatigue: number analyzed (Participants) | 121 | 84
  C12 W89/M23, extreme fatigue | 1 | 0
  C12 W89/M23, fever: number analyzed (Participants) | 121 | 84
  C12 W89/M23, fever | 0 | 0
  C12 W89/M23, night sweats: number analyzed (Participants) | 121 | 84
  C12 W89/M23, night sweats | 3 | 3
  C12 W89/M23, weight loss: number analyzed (Participants) | 121 | 84
  C12 W89/M23, weight loss | 0 | 1
  C13 W97/M25, extreme fatigue: number analyzed (Participants) | 114 | 79
  C13 W97/M25, extreme fatigue | 1 | 0
  C13 W97/M25, fever: number analyzed (Participants) | 114 | 79
  C13 W97/M25, fever | 0 | 0
  C13 W97/M25, night sweats: number analyzed (Participants) | 114 | 79
  C13 W97/M25, night sweats | 2 | 1
  C13 W97/M25, weight loss: number analyzed (Participants) | 114 | 79
  C13 W97/M25, weight loss | 1 | 3
  3M follow up, extreme fatigue: number analyzed (Participants) | 112 | 64
  3M follow up, extreme fatigue | 3 | 2
  3M follow up, fever: number analyzed (Participants) | 112 | 64
  3M follow up, fever | 1 | 1
  3M follow up, night sweats: number analyzed (Participants) | 112 | 64
  3M follow up, night sweats | 4 | 4
  3M follow up, weight loss: number analyzed (Participants) | 112 | 64
  3M follow up, weight loss | 2 | 0
  6M follow up, extreme fatigue: number analyzed (Participants) | 106 | 61
  6M follow up, extreme fatigue | 3 | 2
  6M follow up, fever: number analyzed (Participants) | 106 | 61
  6M follow up, fever | 1 | 0
  6M follow up, night sweats: number analyzed (Participants) | 106 | 61
  6M follow up, night sweats | 2 | 2
  6M follow up, weight loss: number analyzed (Participants) | 106 | 61
  6M follow up, weight loss | 1 | 1
  9M follow up, extreme fatigue: number analyzed (Participants) | 94 | 50
  9M follow up, extreme fatigue | 2 | 2
  9M follow up, fever: number analyzed (Participants) | 94 | 50
  9M follow up, fever | 0 | 0
  9M follow up, night sweats: number analyzed (Participants) | 94 | 50
  9M follow up, night sweats | 4 | 2
  9M follow up, weight loss: number analyzed (Participants) | 94 | 50
  9M follow up, weight loss | 0 | 2
  12M follow up, extreme fatigue: number analyzed (Participants) | 82 | 45
  12M follow up, extreme fatigue | 0 | 3
  12M follow up, fever: number analyzed (Participants) | 82 | 45
  12M follow up, fever | 1 | 1
  12M follow up, night sweats: number analyzed (Participants) | 82 | 45
  12M follow up, night sweats | 2 | 4
  12M follow up, weight loss: number analyzed (Participants) | 82 | 45
  12M follow up, weight loss | 0 | 1
  15M follow up, extreme fatigue: number analyzed (Participants) | 68 | 41
  15M follow up, extreme fatigue | 0 | 0
  15M follow up, fever: number analyzed (Participants) | 68 | 41
  15M follow up, fever | 0 | 1
  15M follow up, night sweats: number analyzed (Participants) | 68 | 41
  15M follow up, night sweats | 2 | 1
  15M follow up, weight loss: number analyzed (Participants) | 68 | 41
  15M follow up, weight loss | 1 | 0
  18M follow up, extreme fatigue: number analyzed (Participants) | 62 | 35
  18M follow up, extreme fatigue | 1 | 1
  18M follow up, fever: number analyzed (Participants) | 62 | 35
  18M follow up, fever | 0 | 0
  18M follow up, night sweats: number analyzed (Participants) | 62 | 35
  18M follow up, night sweats | 2 | 1
  18M follow up, weight loss: number analyzed (Participants) | 62 | 35
  18M follow up, weight loss | 0 | 0
  21M follow up, extreme fatigue: number analyzed (Participants) | 53 | 33
  21M follow up, extreme fatigue | 0 | 1
  21M follow up, fever: number analyzed (Participants) | 53 | 32
  21M follow up, fever | 0 | 0
  21M follow up, night sweats: number analyzed (Participants) | 53 | 32
  21M follow up, night sweats | 1 | 2
  21M follow up, weight loss: number analyzed (Participants) | 53 | 33
  21M follow up, weight loss | 0 | 0
  27M follow up, extreme fatigue: number analyzed (Participants) | 40 | 25
  27M follow up, extreme fatigue | 0 | 0
  27M follow up, fever: number analyzed (Participants) | 40 | 25
  27M follow up, fever | 0 | 0
  27M follow up, night sweats: number analyzed (Participants) | 40 | 24
  27M follow up, night sweats | 2 | 1
  27M follow up, weight loss: number analyzed (Participants) | 40 | 25
  27M follow up, weight loss | 1 | 1
  30M follow up, extreme fatigue: number analyzed (Participants) | 35 | 18
  30M follow up, extreme fatigue | 0 | 0
  30M follow up, fever: number analyzed (Participants) | 35 | 18
  30M follow up, fever | 0 | 0
  30M follow up, night sweats: number analyzed (Participants) | 35 | 18
  30M follow up, night sweats | 1 | 1
  30M follow up, weight loss: number analyzed (Participants) | 35 | 18
  30M follow up, weight loss | 0 | 0
  33M follow up, extreme fatigue: number analyzed (Participants) | 30 | 17
  33M follow up, extreme fatigue | 0 | 0
  33M follow up, fever: number analyzed (Participants) | 30 | 17
  33M follow up, fever | 1 | 0
  33M follow up, night sweats: number analyzed (Participants) | 30 | 17
  33M follow up, night sweats | 2 | 2
  33M follow up, weight loss: number analyzed (Participants) | 30 | 17
  33M follow up, weight loss | 0 | 0
  36M follow up, extreme fatigue: number analyzed (Participants) | 27 | 15
  36M follow up, extreme fatigue | 1 | 0
  36M follow up, fever: number analyzed (Participants) | 27 | 15
  36M follow up, fever | 0 | 0
  36M follow up, night sweats: number analyzed (Participants) | 27 | 15
  36M follow up, night sweats | 1 | 0
  36M follow up, weight loss: number analyzed (Participants) | 27 | 15
  36M follow up, weight loss | 0 | 0
  39M follow up, extreme fatigue: number analyzed (Participants) | 23 | 12
  39M follow up, extreme fatigue | 1 | 0
  39M follow up, fever: number analyzed (Participants) | 23 | 12
  39M follow up, fever | 0 | 0
  39M follow up, night sweats: number analyzed (Participants) | 23 | 12
  39M follow up, night sweats | 1 | 0
  39M follow up, weight loss: number analyzed (Participants) | 23 | 12
  39M follow up, weight loss | 0 | 0
  42M follow up, extreme fatigue: number analyzed (Participants) | 18 | 10
  42M follow up, extreme fatigue | 0 | 0
  42M follow up, fever: number analyzed (Participants) | 18 | 10
  42M follow up, fever | 0 | 1
  42M follow up, night sweats: number analyzed (Participants) | 18 | 10
  42M follow up, night sweats | 0 | 1
  42M follow up,, weight loss: number analyzed (Participants) | 18 | 10
  42M follow up,, weight loss | 0 | 0
  51M follow up, extreme fatigue: number analyzed (Participants) | 8 | 4
  51M follow up, extreme fatigue | 0 | 0
  51M follow up, fever: number analyzed (Participants) | 8 | 4
  51M follow up, fever | 1 | 0
  51M follow up, night sweats: number analyzed (Participants) | 8 | 4
  51M follow up, night sweats | 0 | 1
  51M follow up, weight loss: number analyzed (Participants) | 8 | 4
  51M follow up, weight loss | 0 | 0
  54M follow up, extreme fatigue: number analyzed (Participants) | 6 | 2
  54M follow up, extreme fatigue | 0 | 0
  54M follow up, fever: number analyzed (Participants) | 6 | 2
  54M follow up, fever | 1 | 0
  54M follow up, night sweats: number analyzed (Participants) | 6 | 2
  54M follow up, night sweats | 0 | 0
  54M follow up, weight loss: number analyzed (Participants) | 6 | 2
  54M follow up, weight loss | 0 | 0
  Withdrawal, extreme fatigue: number analyzed (Participants) | 81 | 97
  Withdrawal, extreme fatigue | 9 | 12
  Withdrawal, fever: number analyzed (Participants) | 81 | 97
  Withdrawal, fever | 7 | 3
  Withdrawal, night sweats: number analyzed (Participants) | 81 | 97
  Withdrawal, night sweats | 14 | 15
  Withdrawal, weight loss: number analyzed (Participants) | 81 | 97
  Withdrawal, weight loss | 4 | 10

13. Secondary Outcome: Number of Participants With Grade 3 and Above Adverse Event of Infection
Description: Participants with Grade 3, Grade 4 and Grade 5 adverse event of infection are presented. Adverse events were graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) grade, version 4.0 (1=mild; 2=moderate; 3=severe; 4=life-threatening/disabling; 5=death).
Time Frame: From first dose of study medication until 60 days after the last dose of study medication or until the last observation at Visit 14 (up to 26 months)
Population: Safety Population: all participants who were randomized in the study and analyses were done based on the treatment the participant received regardless of how they were randomized.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 239 | 241
Participants | 38 | 23

14. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From first dose of study medication until 60 days after the last dose of study medication or until the last observation at Visit 14 for AEs (up to 26 months) and until end of study for SAEs (88 months)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 239 | 241
Participants
  Any AE | 221 | 198
  Any SAE | 120 | 120

15. Secondary Outcome: Number of Participants With a Grade 3 or Grade 4 Myelosuppression (Anemia, Neutropenia, or Thrombocytopenia) at Indicated Time Points
Description: Myelosuppression is defined as the decrease in the ability of the bone marrow to produce blood cells. Number of participants who reported myelosuppression (anemia [low hemoglobin count], neutropenia [low neutrophil count], and thrombocytopenia [low platelet count]) are presented. AEs were graded according to NCI common terminology criteria for adverse events (CTCAE) grade, version 4.0 (1, mild; 2, moderate; 3, severe; 4, life-threatening/disabling; 5, death).
Time Frame: From first dose of study medication until 60 days after the last dose of study medication or until the last observation at Visit 14 for AEs (up to 26 months) and until the end of the study for SAEs (88 months)
Population: Safety Population.Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the safety population.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 239 | 241
Participants
  SCR: number analyzed (Participants) | 221 | 199
  SCR | 7 | 5
  C1 W1/M1: number analyzed (Participants) | 3 | 10
  C1 W1/M1 | 1 | 1
  C1 W2/M1: number analyzed (Participants) | 225 | 192
  C1 W2/M1 | 13 | 8
  C2 W9/M3: number analyzed (Participants) | 221 | 210
  C2 W9/M3 | 12 | 15
  C2, unscheduled: number analyzed (Participants) | 5 | 2
  C2, unscheduled | 1 | 0
  C3 W17/M5: number analyzed (Participants) | 208 | 195
  C3 W17/M5 | 18 | 7
  C3, unscheduled: number analyzed (Participants) | 7 | 2
  C3, unscheduled | 1 | 0
  C4 W25/M7: number analyzed (Participants) | 192 | 180
  C4 W25/M7 | 12 | 8
  C4 Unscheduled: number analyzed (Participants) | 1 | 0
  C4 Unscheduled | 1 |
  C5 W33/M9: number analyzed (Participants) | 188 | 164
  C5 W33/M9 | 15 | 5
  C5, unscheduled: number analyzed (Participants) | 3 | 0
  C5, unscheduled | 1 |
  C6 W41/M11: number analyzed (Participants) | 180 | 139
  C6 W41/M11 | 13 | 5
  C6 unscheduled_1: number analyzed (Participants) | 8 | 0
  C6 unscheduled_1 | 4 |
  C6 unscheduled_2: number analyzed (Participants) | 1 | 0
  C6 unscheduled_2 | 1 |
  C7 W49/M13: number analyzed (Participants) | 165 | 132
  C7 W49/M13 | 9 | 2
  C8 W57/M15: number analyzed (Participants) | 148 | 120
  C8 W57/M15 | 10 | 3
  C9 W65/M17: number analyzed (Participants) | 135 | 101
  C9 W65/M17 | 5 | 1
  C9, unscheduled: number analyzed (Participants) | 2 | 1
  C9, unscheduled | 0 | 1
  C10 W73/M19: number analyzed (Participants) | 130 | 101
  C10 W73/M19 | 2 | 2
  C11 W81/M21: number analyzed (Participants) | 122 | 92
  C11 W81/M21 | 5 | 1
  C11 unscheduled_1: number analyzed (Participants) | 2 | 1
  C11 unscheduled_1 | 1 | 0
  C11 unscheduled_2: number analyzed (Participants) | 2 | 0
  C11 unscheduled_2 | 1 |
  C12 W89/M23: number analyzed (Participants) | 115 | 81
  C12 W89/M23 | 3 | 2
  C13 W97/M25: number analyzed (Participants) | 109 | 75
  C13 W97/M25 | 3 | 2
  C13, unscheduled: number analyzed (Participants) | 2 | 0
  C13, unscheduled | 1 |
  3M follow-up: number analyzed (Participants) | 102 | 61
  3M follow-up | 2 | 1
  6M follow-up: number analyzed (Participants) | 92 | 55
  6M follow-up | 2 | 1
  9M follow-up: number analyzed (Participants) | 86 | 50
  9M follow-up | 2 | 1
  12M follow-up: number analyzed (Participants) | 77 | 43
  12M follow-up | 1 | 2
  15M follow-up: number analyzed (Participants) | 62 | 37
  15M follow-up | 1 | 0
  18M follow-up: number analyzed (Participants) | 55 | 33
  18M follow-up | 0 | 1
  27M follow-up: number analyzed (Participants) | 37 | 22
  27M follow-up | 0 | 1
  30M follow-up: number analyzed (Participants) | 29 | 17
  30M follow-up | 0 | 1
  33M follow-up: number analyzed (Participants) | 27 | 16
  33M follow-up | 1 | 0
  60M follow-up: number analyzed (Participants) | 2 | 2
  60M follow-up | 1 | 0
  Withdrawal: number analyzed (Participants) | 76 | 93
  Withdrawal | 11 | 8
  Unscheduled_1: number analyzed (Participants) | 2 | 2
  Unscheduled_1 | 0 | 1
  Unscheduled_2: number analyzed (Participants) | 2 | 5
  Unscheduled_2 | 0 | 2
  Unscheduled_3: number analyzed (Participants) | 7 | 7
  Unscheduled_3 | 1 | 0

16. Secondary Outcome: Number of Participants Who Received at Least One Transfusion During the Study
Description: Participants who received at least one transfusion (any blood products or blood supportive care product) during the study are presented.
Time Frame: From randomization until the end of the study (up to 88 months)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 239 | 241
Participants | 96 | 64

17. Secondary Outcome: Number of Participants Diagnosed With Autoimmune Hemolytic Anemia (AIHA)
Description: AIHA is a disease where the body's immune system fails to recognize red blood cells as "self" and begins destroying these red blood cells. The number of participants diagnosed with AIHA are presented.
Time Frame: From randomization until the end of the study (up to 88 months)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 239 | 241
Participants
  Haemolytic anaemia | 2 | 2
  Autoimmune haemolytic anaemia | 1 | 4
  Thrombocytopenic purpura | 0 | 1

18. Secondary Outcome: Number of Participants With a Positive Anti-ofatumumab Antibody (Human Anti-human Antibody; HAHA) Result
Description: All serum samples for analysis of HAHA were first tested in a screening step; positive samples from the screening were further evaluated in a confirmation test. The confirmed positive samples were reported as HAHA positive and further evaluated in the titration test to obtain a titer of HAHA. A confirmed positive result at any time point means the participant is positive for HAHA.Results are reported as the number of participants positive for HAHA.
Time Frame: Pre-dose (Visit 1), Months 7, 13, 19, and 25 during treatment and at 3 and 6 months after last ofatumumab dose (up to 30 months)
Population: Safety Population. Only those participants with post-ofatumumab HAHA results were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 239 | 0
Participants | 1 |

19. Secondary Outcome: Mean Change From Baseline in the Immunoglobulin (Ig) Antibodies IgA, IgG, and IgM at Indicated Time Points
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Low levels indicate immuno-suppression. IgA, IgG, and IgM were measured in the blood samples of the participants. Baseline IgA, IgG, and IgM values are the last pre-dose assessment values performed on Cycle 1 Day 1. Change from Baseline was calculated as the post-baseline value minus the Baseline value.
Time Frame: Baseline, every six months during treatment, and after last treatment visit and/or upon relapse (up to 88 months)
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the safety population.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 239 | 241
grams per liter
  IgA, C2 W9, M3: number analyzed (Participants) | 0 | 2
  IgA, C2 W9, M3 |  | 0.2 (0.23)
  IgA, C3 W17, M5: number analyzed (Participants) | 6 | 3
  IgA, C3 W17, M5 | 0.0 (0.12) | -0.1 (0.24)
  IgA, C4 W25, M7: number analyzed (Participants) | 189 | 172
  IgA, C4 W25, M7 | -0.1 (0.17) | -0.0 (0.41)
  IgA, C5 W33, M9: number analyzed (Participants) | 1 | 2
  IgA, C5 W33, M9 | -0.0 (NA) — No data was available due to 0 or only 1 participant analyzed. | -0.0 (0.01)
  IgA, C6 W41, M11: number analyzed (Participants) | 1 | 1
  IgA, C6 W41, M11 | 0.0 (NA) — No data was available due to 0 or only 1 participant analyzed. | -0.1 (NA) — No data was available due to 0 or only 1 participant analyzed.
  IgA, C7 W49, M13: number analyzed (Participants) | 157 | 122
  IgA, C7 W49, M13 | -0.1 (0.24) | -0.0 (0.63)
  IgA, C8 W57, M15: number analyzed (Participants) | 3 | 2
  IgA, C8 W57, M15 | -0.1 (0.15) | 0.0 (0.02)
  IgA, C9 W65, M17: number analyzed (Participants) | 3 | 2
  IgA, C9 W65, M17 | -0.2 (0.17) | 0.1 (0.04)
  IgA, C10 W73, M19: number analyzed (Participants) | 125 | 91
  IgA, C10 W73, M19 | -0.1 (0.20) | 0.1 (0.37)
  IgA, C11 W81, M21: number analyzed (Participants) | 1 | 2
  IgA, C11 W81, M21 | -0.0 (NA) — No data was available due to 0 or only 1 participant analyzed. | 0.2 (0.21)
  IgA, C12 W89, M23: number analyzed (Participants) | 1 | 4
  IgA, C12 W89, M23 | -0.3 (NA) — No data was available due to 0 or only 1 participant analyzed. | 0.2 (0.39)
  IgA, C13 W97, M25: number analyzed (Participants) | 107 | 74
  IgA, C13 W97, M25 | -0.1 (0.23) | 0.1 (0.38)
  IgA, 3M FU: number analyzed (Participants) | 89 | 51
  IgA, 3M FU | -0.1 (0.22) | 0.2 (0.37)
  IgA, 6M FU: number analyzed (Participants) | 83 | 50
  IgA, 6M FU | -0.1 (0.18) | 0.1 (0.39)
  IgA, 9M FU: number analyzed (Participants) | 62 | 40
  IgA, 9M FU | -0.1 (0.22) | 0.1 (0.38)
  IgA, 12M FU: number analyzed (Participants) | 54 | 35
  IgA, 12M FU | -0.1 (0.30) | 0.2 (0.36)
  IgA, 15M FU: number analyzed (Participants) | 40 | 31
  IgA, 15M FU | -0.0 (0.27) | 0.2 (0.44)
  IgA, 18M FU: number analyzed (Participants) | 38 | 23
  IgA, 18M FU | 0.1 (0.57) | 0.1 (0.25)
  IgA, 21M FU: number analyzed (Participants) | 33 | 23
  IgA, 21M FU | -0.1 (0.40) | 0.1 (0.34)
  IgA, 24M FU: number analyzed (Participants) | 29 | 21
  IgA, 24M FU | 0.2 (1.06) | 0.1 (0.37)
  IgA, 27M FU: number analyzed (Participants) | 24 | 15
  IgA, 27M FU | 0.1 (0.70) | 0.1 (0.46)
  IgA, 30M FU: number analyzed (Participants) | 18 | 12
  IgA, 30M FU | 0.2 (0.85) | 0.1 (0.58)
  IgA, 33M FU: number analyzed (Participants) | 18 | 11
  IgA, 33M FU | 0.4 (1.48) | 0.2 (0.60)
  IgA, 36M FU: number analyzed (Participants) | 18 | 11
  IgA, 36M FU | 0.2 (1.06) | 0.2 (0.63)
  IgA, 39M FU: number analyzed (Participants) | 14 | 8
  IgA, 39M FU | 0.2 (0.86) | 0.3 (0.71)
  IgA, 42M FU: number analyzed (Participants) | 14 | 6
  IgA, 42M FU | 0.4 (1.67) | 0.2 (0.72)
  IgA, 45M FU: number analyzed (Participants) | 11 | 4
  IgA, 45M FU | -0.2 (0.20) | 0.4 (0.94)
  IgA, 48M FU: number analyzed (Participants) | 9 | 3
  IgA, 48M FU | -0.1 (0.83) | -0.0 (0.25)
  IgA, 51M FU: number analyzed (Participants) | 4 | 3
  IgA, 51M FU | 0.3 (1.15) | 0.2 (0.70)
  IgA, 54M FU: number analyzed (Participants) | 6 | 2
  IgA, 54M FU | 0.0 (0.89) | 0.7 (1.34)
  IgA, 57M FU: number analyzed (Participants) | 3 | 2
  IgA, 57M FU | -0.4 (0.36) | 0.4 (1.04)
  IgA, 60M FU: number analyzed (Participants) | 2 | 2
  IgA, 60M FU | -0.5 (0.42) | 0.4 (1.05)
  IgA, Withdrawal: number analyzed (Participants) | 6 | 4
  IgA, Withdrawal | 0.0 (0.53) | -0.1 (0.08)
  IgG, C2 W9, M3: number analyzed (Participants) | 0 | 2
  IgG, C2 W9, M3 |  | -0.4 (0.21)
  IgG, C3 W17, M5: number analyzed (Participants) | 6 | 3
  IgG, C3 W17, M5 | 0.0 (1.17) | 0.2 (0.39)
  IgG, C4 W25, M7: number analyzed (Participants) | 190 | 172
  IgG, C4 W25, M7 | -0.7 (2.03) | -0.1 (1.83)
  IgG, C5 W33, M9: number analyzed (Participants) | 1 | 2
  IgG, C5 W33, M9 | -1.0 (NA) — No data was available due to 0 or only 1 participant analyzed. | 0.5 (2.20)
  IgG, C6 W41, M11: number analyzed (Participants) | 1 | 1
  IgG, C6 W41, M11 | -1.9 (NA) — No data was available due to 0 or only 1 participant analyzed. | 1.0 (NA) — No data was available due to 0 or only 1 participant analyzed.
  IgG, C7 W49, M13: number analyzed (Participants) | 157 | 122
  IgG, C7 W49, M13 | -1.1 (1.9) | 0.2 (2.88)
  IgG, C8 W57, M15: number analyzed (Participants) | 3 | 2
  IgG, C8 W57, M15 | -1.3 (1.03) | -0.9 (0.08)
  IgG, C9 W65, M17: number analyzed (Participants) | 3 | 2
  IgG, C9 W65, M17 | -3.7 (4.96) | 0.9 (0.71)
  IgG, C10 W73, M19: number analyzed (Participants) | 125 | 91
  IgG, C10 W73, M19 | -1.0 (2.15) | 0.6 (4.61)
  IgG, C11 W81, M21: number analyzed (Participants) | 1 | 2
  IgG, C11 W81, M21 | 0.2 (NA) — No data was available due to 0 or only 1 participant analyzed. | -0.3 (1.39)
  IgG, C12 W89, M23: number analyzed (Participants) | 1 | 4
  IgG, C12 W89, M23 | -0.5 (NA) — No data was available due to 0 or only 1 participant analyzed. | 0.2 (0.89)
  IgG, C13 W97, M25: number analyzed (Participants) | 107 | 74
  IgG, C13 W97, M25 | -1.1 (2.45) | 0.3 (3.02)
  IgG, 3M FU: number analyzed (Participants) | 90 | 51
  IgG, 3M FU | -0.7 (2.46) | 0.2 (2.83)
  IgG, 6M FU: number analyzed (Participants) | 83 | 50
  IgG, 6M FU | -0.9 (2.24) | 0.2 (2.89)
  IgG, 9M FU: number analyzed (Participants) | 62 | 40
  IgG, 9M FU | -0.7 (2.29) | 0.1 (2.87)
  IgG, 12M FU: number analyzed (Participants) | 54 | 35
  IgG, 12M FU | -0.5 (2.17) | -0.3 (3.26)
  IgG, 15M FU: number analyzed (Participants) | 40 | 31
  IgG, 15M FU | -0.4 (2.49) | -0.1 (3.29)
  IgG, 18M FU: number analyzed (Participants) | 38 | 23
  IgG, 18M FU | -0.5 (2.71) | -0.3 (3.45)
  IgG, 21M FU: number analyzed (Participants) | 33 | 23
  IgG, 21M FU | -0.9 (2.39) | 0.1 (3.81)
  IgG, 24M FU (: number analyzed (Participants) | 29 | 21
  IgG, 24M FU ( | -0.1 (2.17) | 0.0 (3.43)
  IgG, 27M FU: number analyzed (Participants) | 24 | 15
  IgG, 27M FU | -0.3 (2.32) | -0.5 (3.97)
  IgG, 30M FU: number analyzed (Participants) | 18 | 12
  IgG, 30M FU | 0.3 (2.67) | -0.9 (4.83)
  IgG, 33M FU: number analyzed (Participants) | 18 | 11
  IgG, 33M FU | 0.7 (2.91) | -1.1 (5.63)
  IgG, 36M FU: number analyzed (Participants) | 18 | 11
  IgG, 36M FU | -0.1 (2.71) | -1.2 (3.87)
  IgG, 39M FU: number analyzed (Participants) | 14 | 8
  IgG, 39M FU | 0.3 (2.53) | -0.9 (5.60)
  IgG, 42M FU: number analyzed (Participants) | 14 | 6
  IgG, 42M FU | 0.6 (3.03) | 0.9 (4.82)
  IgG, 45M FU: number analyzed (Participants) | 11 | 4
  IgG, 45M FU | -0.6 (2.11) | 2.3 (4.00)
  IgG, 48M FU: number analyzed (Participants) | 9 | 3
  IgG, 48M FU | -0.6 (2.30) | 3.5 (3.14)
  IgG, 51M FU: number analyzed (Participants) | 4 | 3
  IgG, 51M FU | 0.1 (3.25) | 2.4 (4.02)
  IgG, 54M FU: number analyzed (Participants) | 6 | 2
  IgG, 54M FU | -1.0 (2.35) | 5.6 (4.14)
  IgG, 57M FU: number analyzed (Participants) | 3 | 2
  IgG, 57M FU | 1.3 (4.01) | 5.3 (5.68)
  IgG, 60M FU: number analyzed (Participants) | 2 | 2
  IgG, 60M FU | 0.8 (4.43) | 4.6 (4.28)
  IgG, Withdrawal: number analyzed (Participants) | 6 | 4
  IgG, Withdrawal | -0.7 (0.91) | -1.5 (1.86)
  IgM, C2 W9, M3: number analyzed (Participants) | 0 | 2
  IgM, C2 W9, M3 |  | 0.1 (0.12)
  IgM, C3 W17, M5: number analyzed (Participants) | 6 | 3
  IgM, C3 W17, M5 | -0.0 (0.09) | -0.0 (0.06)
  IgM, C4 W25, M7: number analyzed (Participants) | 190 | 172
  IgM, C4 W25, M7 | -0.1 (0.43) | 0.1 (0.42)
  IgM, C5 W33, M9: number analyzed (Participants) | 1 | 2
  IgM, C5 W33, M9 | -0.1 (NA) — No data was available due to 0 or only 1 participant analyzed. | -0.1 (0.07)
  IgM, C6 W41, M11: number analyzed (Participants) | 1 | 1
  IgM, C6 W41, M11 | -0.5 (NA) — No data was available due to 0 or only 1 participant analyzed. | 0.0 (NA) — No data was available due to 0 or only 1 participant analyzed.
  IgM, C7 W49, M13: number analyzed (Participants) | 157 | 122
  IgM, C7 W49, M13 | -0.1 (0.29) | 0.2 (0.90)
  IgM, C8 W57, M15: number analyzed (Participants) | 3 | 2
  IgM, C8 W57, M15 | -0.0 (0.05) | -0.0 (0.01)
  IgM, C9 W65, M17: number analyzed (Participants) | 3 | 2
  IgM, C9 W65, M17 | -0.3 (0.54) | 0.3 (0.49)
  IgM, C10 W73, M19: number analyzed (Participants) | 125 | 91
  IgM, C10 W73, M19 | -0.1 (0.36) | 0.2 (0.86)
  IgM, C11 W81, M21: number analyzed (Participants) | 1 | 2
  IgM, C11 W81, M21 | 0.0 (NA) — No data was available due to 0 or only 1 participant analyzed. | 0.2 (0.04)
  IgM, C12 W89, M23: number analyzed (Participants) | 1 | 4
  IgM, C12 W89, M23 | 0.0 (NA) — No data was available due to 0 or only 1 participant analyzed. | -0.0 (0.11)
  IgM, C13 W97, M25: number analyzed (Participants) | 107 | 74
  IgM, C13 W97, M25 | -0.1 (0.45) | 0.2 (0.79)
  IgM, 3M FU: number analyzed (Participants) | 90 | 51
  IgM, 3M FU | -0.0 (0.35) | 0.3 (1.30)
  IgM, 6M FU (: number analyzed (Participants) | 83 | 50
  IgM, 6M FU ( | -0.1 (0.36) | 0.4 (1.60)
  IgM, 9M FU: number analyzed (Participants) | 62 | 40
  IgM, 9M FU | -0.1 (0.17) | 0.6 (2.93)
  IgM, 12M FU: number analyzed (Participants) | 54 | 35
  IgM, 12M FU | -0.0 (0.18) | 0.6 (2.49)
  IgM, 15M FU: number analyzed (Participants) | 40 | 31
  IgM, 15M FU | -0.0 (0.15) | 0.3 (1.08)
  IgM, 18M FU: number analyzed (Participants) | 38 | 23
  IgM, 18M FU | 0.1 (0.25) | 1.2 (4.95)
  IgM, 21M FU: number analyzed (Participants) | 33 | 23
  IgM, 21M FU | 0.1 (0.41) | 1.4 (5.48)
  IgM, 24M FU: number analyzed (Participants) | 29 | 21
  IgM, 24M FU | 0.0 (0.14) | 2.0 (8.19)
  IgM, 27M FU: number analyzed (Participants) | 24 | 15
  IgM, 27M FU | 0.2 (0.41) | -0.2 (1.14)
  IgM, 30M FU (n=18, 12): number analyzed (Participants) | 18 | 12
  IgM, 30M FU (n=18, 12) | 0.1 (0.17) | -0.0 (1.51)
  IgM, 33M FU: number analyzed (Participants) | 18 | 11
  IgM, 33M FU | 0.1 (0.22) | 0.1 (0.36)
  IgM, 36M FU: number analyzed (Participants) | 18 | 11
  IgM, 36M FU | 0.2 (0.28) | -0.3 (1.31)
  IgM, 39M FU: number analyzed (Participants) | 14 | 8
  IgM, 39M FU | 0.1 (0.21) | -0.4 (1.54)
  IgM, 42M FU: number analyzed (Participants) | 14 | 6
  IgM, 42M FU | 0.1 (0.23) | -0.6 (1.79)
  IgM, 45M FU: number analyzed (Participants) | 11 | 4
  IgM, 45M FU | 0.2 (0.32) | 0.2 (0.27)
  IgM, 48M FU: number analyzed (Participants) | 9 | 3
  IgM, 48M FU | 0.1 (0.28) | 0.4 (0.38)
  IgM, 51M FU: number analyzed (Participants) | 4 | 3
  IgM, 51M FU | -0.0 (0.06) | 0.3 (0.39)
  IgM, 54M FU: number analyzed (Participants) | 6 | 2
  IgM, 54M FU | 0.1 (0.24) | 0.5 (0.26)
  IgM, 57M FU: number analyzed (Participants) | 3 | 2
  IgM, 57M FU | 0.2 (0.49) | 0.4 (0.41)
  IgM, 60M FU: number analyzed (Participants) | 2 | 2
  IgM, 60M FU | 0.6 (0.84) | 0.4 (0.42)
  IgM, Withdrawal: number analyzed (Participants) | 6 | 4
  IgM, Withdrawal | 0.3 (0.73) | -0.0 (0.03)

20. Secondary Outcome: Number of Participants Who Were Positive and Negative for Minimal Residual Disease (MRD) at Any Visit
Description: MRD refers to small number of leukemic cells that remain in the participant during treatment or after treatment at the time the participant achieved a confirmed complete remission. Number of participants who were positive and negative for minimal residual disease (MRD) at any visit is presented.
Time Frame: From randomization until the end of the study (up to 88 months)
Population: ITT Population. Only those participants with data available at the specified time point were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 240 | 240
Participants
  Positive: number analyzed (Participants) | 177 | 159
  Positive | 150 | 122
  Negative: number analyzed (Participants) | 177 | 159
  Negative | 27 | 37

21. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD) CD5+CD19+ and CD5-CD19+ Cell Counts at the Indicated Time Points
Description: CD5+CD19+ cells were counted by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus. Baseline CD5+CD19+ and CD5-CD19+ cell count value is the last pre-dose assessment values performed on Cycle 1 Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and every two months from Month 3 until Month 25 and at every followup (up to 88 months)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 240 | 240
Cells per microliter
  CD5+CD19+, C2 W9, M3: number analyzed (Participants) | 192 | 166
  CD5+CD19+, C2 W9, M3 | -284.1 (2101.26) | 598.6 (3155.69)
  CD5+CD19+, C3 W17, M5: number analyzed (Participants) | 185 | 169
  CD5+CD19+, C3 W17, M5 | 52.0 (3554.94) | 750.5 (1995.47)
  CD5+CD19+, C4 W25, M7: number analyzed (Participants) | 170 | 152
  CD5+CD19+, C4 W25, M7 | -177.6 (4105.41) | 2102.2 (9866.31)
  CD5+CD19+, C5 W33, M9: number analyzed (Participants) | 168 | 147
  CD5+CD19+, C5 W33, M9 | -113.6 (3336.44) | 1905.2 (6104.84)
  CD5+CD19+, C6 W41, M11: number analyzed (Participants) | 154 | 129
  CD5+CD19+, C6 W41, M11 | -450.3 (2851.41) | 1550.9 (5483.76)
  CD5+CD19+, C7 W49, M13: number analyzed (Participants) | 152 | 122
  CD5+CD19+, C7 W49, M13 | -505.3 (2716.66) | 1429.2 (4408.69)
  CD5+CD19+, C8 W57, M15: number analyzed (Participants) | 137 | 108
  CD5+CD19+, C8 W57, M15 | -625.9 (3003.35) | 1107.6 (3371.04)
  CD5+CD19+, C9 W65, M17: number analyzed (Participants) | 123 | 90
  CD5+CD19+, C9 W65, M17 | -649.5 (3057.32) | 967.0 (1826.90)
  CD5+CD19+, C10 W73, M19: number analyzed (Participants) | 120 | 89
  CD5+CD19+, C10 W73, M19 | -238.6 (4061.13) | 1146.0 (1914.02)
  CD5+CD19+, C11 W81, M21: number analyzed (Participants) | 112 | 89
  CD5+CD19+, C11 W81, M21 | -579.0 (3446.95) | 1656.7 (2662.28)
  CD5+CD19+, C12 W89, M23: number analyzed (Participants) | 110 | 74
  CD5+CD19+, C12 W89, M23 | -569.5 (3510.43) | 1608.3 (3220.20)
  CD5+CD19+, C13 W97, M25: number analyzed (Participants) | 100 | 64
  CD5+CD19+, C13 W97, M25 | -361.3 (2702.79) | 2059.0 (4987.97)
  CD5+CD19+, 3M FU: number analyzed (Participants) | 92 | 53
  CD5+CD19+, 3M FU | 121.1 (5479.03) | 2143.9 (4280.66)
  CD5+CD19+, 6M FU: number analyzed (Participants) | 89 | 48
  CD5+CD19+, 6M FU | 1968.3 (15975.52) | 2363.5 (4937.00)
  CD5+CD19+, 9M FU: number analyzed (Participants) | 82 | 41
  CD5+CD19+, 9M FU | 1411.3 (6965.41) | 4008.5 (13550.03)
  CD5+CD19+, 12M FU: number analyzed (Participants) | 74 | 35
  CD5+CD19+, 12M FU | 2198.5 (10743.58) | 2316.0 (8763.12)
  CD5+CD19+, 15M FU: number analyzed (Participants) | 57 | 30
  CD5+CD19+, 15M FU | -84.4 (4140.77) | 1246.2 (2894.20)
  CD5+CD19+, 18M FU: number analyzed (Participants) | 48 | 27
  CD5+CD19+, 18M FU | 1844.1 (10091.28) | 1250.9 (3182.14)
  CD5+CD19+, 21M FU: number analyzed (Participants) | 42 | 24
  CD5+CD19+, 21M FU | -395.1 (4521.30) | 1147.5 (2191.69)
  CD5+CD19+, 24M FU: number analyzed (Participants) | 38 | 24
  CD5+CD19+, 24M FU | 279.4 (6250.23) | 2354.0 (6726.31)
  CD5+CD19+, 27M FU: number analyzed (Participants) | 34 | 20
  CD5+CD19+, 27M FU | -368.6 (4829.16) | 2250.8 (5833.72)
  CD5+CD19+, 30M FU: number analyzed (Participants) | 27 | 16
  CD5+CD19+, 30M FU | -354.4 (5686.14) | 2189.3 (6246.05)
  CD5+CD19+, 33M FU: number analyzed (Participants) | 23 | 14
  CD5+CD19+, 33M FU | -397.0 (2767.27) | 3024.8 (7543.26)
  CD5+CD19+, 36M FU: number analyzed (Participants) | 23 | 13
  CD5+CD19+, 36M FU | -354.8 (2767.77) | 3668.4 (8581.98)
  CD5+CD19+, 39M FU: number analyzed (Participants) | 19 | 10
  CD5+CD19+, 39M FU | -163.7 (3116.92) | 1217.1 (2441.59)
  CD5+CD19+, 42M FU: number analyzed (Participants) | 16 | 9
  CD5+CD19+, 42M FU | -81.7 (3426.53) | 2005.9 (4327.53)
  CD5+CD19+, 45M FU: number analyzed (Participants) | 13 | 7
  CD5+CD19+, 45M FU | 466.9 (919.60) | 450.4 (1031.86)
  CD5+CD19+, 48M FU: number analyzed (Participants) | 10 | 5
  CD5+CD19+, 48M FU | 1255.3 (2289.34) | 643.4 (1270.16)
  CD5+CD19+, 51M FU: number analyzed (Participants) | 5 | 4
  CD5+CD19+, 51M FU | 4341.4 (8803.05) | 1104.8 (2004.49)
  CD5+CD19+, 54M FU: number analyzed (Participants) | 5 | 2
  CD5+CD19+, 54M FU | 1689.8 (2357.27) | 237.5 (251.02)
  CD5+CD19+, 57M FU: number analyzed (Participants) | 3 | 2
  CD5+CD19+, 57M FU | 703.3 (898.82) | 186.0 (145.66)
  CD5+CD19+, 60M FU: number analyzed (Participants) | 2 | 2
  CD5+CD19+, 60M FU | 237.0 (326.68) | 278.5 (392.44)
  CD5+CD19+, withdrawal: number analyzed (Participants) | 73 | 83
  CD5+CD19+, withdrawal | 8916.4 (25922.35) | 13991.9 (23553.42)
  CD5-CD19+, C2 W9, M3: number analyzed (Participants) | 192 | 166
  CD5-CD19+, C2 W9, M3 | -17.9 (588.42) | 81.1 (781.76)
  CD5-CD19+, C3 W17, M5: number analyzed (Participants) | 185 | 169
  CD5-CD19+, C3 W17, M5 | 5.2 (358.12) | 50.7 (168.87)
  CD5-CD19+, C4 W25, M7: number analyzed (Participants) | 170 | 152
  CD5-CD19+, C4 W25, M7 | 73.9 (687.62) | 228.2 (2037.16)
  CD5-CD19+, C5 W33, M9: number analyzed (Participants) | 168 | 147
  CD5-CD19+, C5 W33, M9 | 87.5 (971.22) | 98.9 (401.27)
  CD5-CD19+, C6 W41, M11: number analyzed (Participants) | 154 | 129
  CD5-CD19+, C6 W41, M11 | -13.1 (257.81) | 92.7 (296.23)
  CD5-CD19+, C7 W49, M13: number analyzed (Participants) | 152 | 122
  CD5-CD19+, C7 W49, M13 | 5.3 (368.66) | 77.5 (125.81)
  CD5-CD19+, C8 W57, M15: number analyzed (Participants) | 137 | 108
  CD5-CD19+, C8 W57, M15 | -13.3 (279.89) | 95.9 (143.95)
  CD5-CD19+, C9 W65, M17: number analyzed (Participants) | 123 | 90
  CD5-CD19+, C9 W65, M17 | -4.4 (349.91) | 128.3 (294.11)
  CD5-CD19+, C10 W73, M19: number analyzed (Participants) | 120 | 89
  CD5-CD19+, C10 W73, M19 | 3.3 (421.97) | 172.5 (555.27)
  CD5-CD19+, C11 W81, M21: number analyzed (Participants) | 112 | 89
  CD5-CD19+, C11 W81, M21 | -20.7 (303.21) | 127.2 (150.18)
  CD5-CD19+, C12 W89, M23: number analyzed (Participants) | 110 | 74
  CD5-CD19+, C12 W89, M23 | -13.5 (306.57) | 143.7 (251.88)
  CD5-CD19+, C13 W97, M25: number analyzed (Participants) | 100 | 64
  CD5-CD19+, C13 W97, M25 | 7.9 (103.85) | 184.0 (403.97)
  CD5-CD19+, 3M FU: number analyzed (Participants) | 92 | 53
  CD5-CD19+, 3M FU | 27.4 (522.67) | 145.7 (229.93)
  CD5-CD19+, 6M FU: number analyzed (Participants) | 89 | 48
  CD5-CD19+, 6M FU | 22.6 (428.70) | 153.8 (330.63)
  CD5-CD19+, 9M FU: number analyzed (Participants) | 82 | 41
  CD5-CD19+, 9M FU | 13.2 (368.63) | 140.9 (107.92)
  CD5-CD19+, 12M FU: number analyzed (Participants) | 74 | 35
  CD5-CD19+, 12M FU | 86.4 (769.73) | 147.2 (136.93)
  CD5-CD19+, 15M FU: number analyzed (Participants) | 57 | 30
  CD5-CD19+, 15M FU | 10.8 (393.47) | 154.8 (120.86)
  CD5-CD19+, 18M FU: number analyzed (Participants) | 48 | 27
  CD5-CD19+, 18M FU | 84.7 (146.38) | 173.5 (142.95)
  CD5-CD19+, 21M FU: number analyzed (Participants) | 42 | 24
  CD5-CD19+, 21M FU | 16.2 (450.95) | 175.9 (158.31)
  CD5-CD19+, 24M FU: number analyzed (Participants) | 38 | 24
  CD5-CD19+, 24M FU | 574.7 (2993.58) | 223.2 (200.06)
  CD5-CD19+, 27M FU: number analyzed (Participants) | 34 | 20
  CD5-CD19+, 27M FU | 102.0 (643.44) | 153.3 (110.37)
  CD5-CD19+, 30M FU: number analyzed (Participants) | 27 | 16
  CD5-CD19+, 30M FU | 38.7 (271.84) | 142.9 (106.57)
  CD5-CD19+, 33M FU: number analyzed (Participants) | 23 | 14
  CD5-CD19+, 33M FU | 98.3 (117.18) | 157.5 (96.69)
  CD5-CD19+, 36M FU: number analyzed (Participants) | 23 | 13
  CD5-CD19+, 36M FU | 141.1 (179.33) | 215.2 (298.90)
  CD5-CD19+, 39M FU: number analyzed (Participants) | 19 | 10
  CD5-CD19+, 39M FU | 134.3 (167.33) | 183.9 (249.78)
  CD5-CD19+, 42M FU: number analyzed (Participants) | 16 | 9
  CD5-CD19+, 42M FU | 113.3 (131.48) | 361.1 (601.36)
  CD5-CD19+, 45M FU: number analyzed (Participants) | 13 | 7
  CD5-CD19+, 45M FU | 108.6 (140.97) | 157.7 (116.04)
  CD5-CD19+, 48M FU: number analyzed (Participants) | 10 | 5
  CD5-CD19+, 48M FU | 147.7 (185.10) | 180.6 (175.93)
  CD5-CD19+, 51M FU: number analyzed (Participants) | 5 | 4
  CD5-CD19+, 51M FU | 162.6 (229.87) | 139.3 (82.75)
  CD5-CD19+, 54M FU: number analyzed (Participants) | 5 | 2
  CD5-CD19+, 54M FU | 221.2 (217.75) | 315.0 (43.84)
  CD5-CD19+, 57M FU: number analyzed (Participants) | 3 | 2
  CD5-CD19+, 57M FU | 138.3 (196.32) | 195.5 (17.68)
  CD5-CD19+, 60M FU: number analyzed (Participants) | 2 | 2
  CD5-CD19+, 60M FU | 180.5 (222.74) | 127.0 (173.95)
  CD5-CD19+, withdrawal: number analyzed (Participants) | 73 | 83
  CD5-CD19+, withdrawal | 593.5 (2028.89) | 552.7 (1799.49)

22. Secondary Outcome: Summary of Covariates to Compute Cox Proportional Hazards Regression Model for Relationship Between Investigator Assessed Progression-free Survival and the Indicated Prognostic Markers
Description: Blood samples were collected for the assessment of the following prognostic markers at Baseline (BL) and upon relapse: immunoglobulin heavy chain variable region (IgVH) mutational status; VH3-21 usage; Cytogenetics (by fluorescent in situ hybridization [FISH]) including 6q-, 11q-, +12q, 17p-, 13q- deletions; beta 2 microglobulin. Cox-regression model was used to explore the relationship between progression-free survival and the following explanatory variables: treatment group, cytogenetics (analyzed by FISH) at BL, IgVH mutational status at BL, beta 2 microglobulin at BL, BL CD20 and BL complement level. For each covariate, a hazard ratio <1 indicates a lower risk on the first effect tested compared with the other effects tested. Cytogenetics Group (based on >=20%)=CY G.
Time Frame: From Baseline until the end of the study (up to 79 months)
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 240 | 240
Participants
  CY G: 6q- or +12q or 13q | 36 | 12
  CY G: 17p- | 7 | 4
  CY G: 11q- | 11 | 10
  CY G: no aberration | 166 | 181
  CY G: missing | 20 | 33
  B2 Microglobulin G 2: > 3500 μg/L | 80 | 68
  B2 Microglobulin G 2: <=3500 μg/L | 157 | 171
  B2 Microglobulin G 2: missing | 3 | 1
  IgVH Mutational Status 1: mutated | 54 | 74
  IgVH Mutational Status 1: unmutated | 139 | 116
  IgVH Mutational Status 1: not available | 3 | 1
  IgVH Mutational Status 1: missing | 44 | 49
  VH3-21 Usage Flag: Yes | 7 | 7
  VH3-21 Usage Flag: No | 233 | 233
Statistical Analysis 1: Comparison: Ofatumumab; Test type: Superiority; Hazard Ratio (HR) = 1.547, 95% CI 2-sided [1.051 to 2.276] — HR estimated for Cytogenetics Group (based on >=20% cut-off) with 6q-, or +12q or 13q-/no abberation
Statistical Analysis 2: Comparison: Ofatumumab; Test type: Superiority; Hazard Ratio (HR) = 9.303, 95% CI 2-sided [4.934 to 17.540] — HR estimated for Cytogenetics Group (based on >=20% cut-off) with 17p-/no abberation
Statistical Analysis 3: Comparison: Ofatumumab; Test type: Superiority; Hazard Ratio (HR) = 4.219, 95% CI 2-sided [2.468 to 7.210] — HR estimated for Cytogenetics Group (based on >=20% cut-off) with 11q-/no abberation
Statistical Analysis 4: Comparison: Ofatumumab; Test type: Superiority; Hazard Ratio (HR) = 1.832, 95% CI 2-sided [1.434 to 2.339] — HR estimated for B2 Microglobulin Group 2 with 3500 as cut off: >3500 ug/L/<=3500 ug/L
Statistical Analysis 5: Comparison: Ofatumumab; Test type: Superiority; Hazard Ratio (HR) = 0.573, 95% CI 2-sided [0.432 to 0.760] — HR estimated for IgVH Mutational Status 1 Mutated/Unmutated
Statistical Analysis 6: Comparison: Ofatumumab; Test type: Superiority; Hazard Ratio (HR) = 1.301, 95% CI 2-sided [0.692 to 2.448] — HR estimated for VH3-21 Usage Flag Yes/No

23. Secondary Outcome: Cmax and Ctrough of Ofatumumab
Description: Blood samples were collected to assess the plasma concentration of ofatumumab. Maximum concentration (Cmax) and observed drug concentration prior to the next dose (Ctrough) were determined. Blood samples were collected at pre-dose and 0.5 hours after the end of the infusion at treatment on Month 1 Week 1 (Day 1), Month 1 Week 2 (Day 8), and at every second infusion.
Time Frame: Day 1 of Month 1 (Cycle 1 Week 1); Day 8 of Month 1 (Cycle 1 Week 2); and Month 7 (Cycle 4)
Population: Pharmacokinetic (PK) Population: all participants in the ITT Population for whom a PK sample was obtained and analyzed. Only those participants available at the indicated time points (indicated by n=X in the category titles) were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 221 | 0
micrograms per milliliter (µg/mL)
  Cmax, Cycle 1 Week 1: number analyzed (Participants) | 219 | 0
  Cmax, Cycle 1 Week 1 | 73.8 (65) |
  Cmax, Cycle 1 Week 2: number analyzed (Participants) | 212 | 0
  Cmax, Cycle 1 Week 2 | 264 (50) |
  Cmax, Cycle 4: number analyzed (Participants) | 157 | 0
  Cmax, Cycle 4 | 275 (31) |
  Ctrough, Cycle 1 Week 2: number analyzed (Participants) | 218 | 0
  Ctrough, Cycle 1 Week 2 | 16.3 (254) |
  Ctrough, Cycle 4: number analyzed (Participants) | 164 | 0
  Ctrough, Cycle 4 | 9.9 (1323) |

24. Secondary Outcome: Total Plasma Clearance (CL) of Ofatumumab
Description: Plasma clearance is defined as the plasma volume that is cleared of drug per unit of time.
Time Frame: Day 1 of Month 1 (Cycle 1 Week 1); Day 8 of Month 1 (Cycle 1 Week 2); and Month 7 (Cycle 4)
Population: PK Population. Only those participants available at the indicated time points (indicated by n=X in the category titles) were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millileters per hour (mL/hour)
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 190 | 0
millileters per hour (mL/hour)
  Cycle 1 Week 1 | 49.1 (38) |
  Cycle 1 Week 2: number analyzed (Participants) | 173 | 0
  Cycle 1 Week 2 | 9.6 (43) |
  Cycle 4: number analyzed (Participants) | 124 | 0
  Cycle 4 | 8.1 (50) |

25. Secondary Outcome: AUC(0-tau) of Ofatumumab
Description: Area under the concentration time curve over the dosing interval (AUC[0-tau]) is a measure of the drug exposure over time.
Time Frame: Day 1 of Month 1 (Cycle 1 Week 1); Day 8 of Month 1 (Cycle 1 Week 2); and Month 7 (Cycle 4)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per mL (µg*hour/mL)
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 190 | 0
micrograms*hour per mL (µg*hour/mL)
  Cycle 1 Week 1 | 6113 (38) |
  Cycle 1 Week 2: number analyzed (Participants) | 173 | 0
  Cycle 1 Week 2 | 104013 (43) |
  Cycle 4: number analyzed (Participants) | 124 | 0
  Cycle 4 | 122782 (50) |

26. Secondary Outcome: Vss of Ofatumumab
Description: Volume of distribution at steady state (Vss) is defined as the apparent volume of distribution of a drug between plasma and the rest of the body at steady state. Data from all time points collected were used to calculate one Vss value for each individual.
Time Frame: Day 1 Month 1 ( Cycle 1) through Month 7 ( Cycle 4)
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 224 | 0
Liters (L) | 6.0 (27) |

27. Secondary Outcome: Plasma Half-life (t1/2) of Ofatumumab
Description: The terminal half life (t1/2) of ofatumumab is defined as the time required for the plasma concentration of ofatumumab to reach half of its original value.
Time Frame: Day 1 of Month 1 (Cycle 1 Week 1); Day 8 of Month 1 (Cycle 1 Week 2); and Month 7 (Cycle 4)
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Ofatumumab | Observation
Number analyzed (Participants) | 190 | 0
hours
  Cycle 1 Week 1 | 126 (35) |
  Cycle 1 Week 2: number analyzed (Participants) | 173 | 0
  Cycle 1 Week 2 | 458 (36) |
  Cycle 4: number analyzed (Participants) | 124 | 0
  Cycle 4 | 542 (48) |

ADVERSE EVENTS:
Time Frame: From first dose of study medication until 60 days after the last dose of study medication or until the last observation at Visit 14 for AEs (up to 26 months) and until end of study for SAEs (88 months).
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of 88 months.
Groups:
- Total: All patients
Arm/Group | Ofatumumab | Observation | Total
All-Cause Mortality (participants affected / at risk) | 88/239 | 87/241 | 175/480
Serious Adverse Events (participants affected / at risk) | 120/239 | 120/241 | 240/480
Other Adverse Events (participants affected / at risk) | 202/239 | 139/241 | 341/480
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=239) | Observation (N=241) | Total (N=480)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 7 | 12
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 18 | 10 | 28
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 1 | 3
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 5 | 10
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 4
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 4
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2 | 3
Cardiac failure (Cardiac disorders) | 3 | 2 | 5
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 3 | 4
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 1 | 2
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0 | 2
Eosinophilic colitis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 2
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Chest pain (General disorders) | 0 | 2 | 2
Condition aggravated (General disorders) | 0 | 1 | 1
General physical health deterioration (General disorders) | 4 | 3 | 7
Malaise (General disorders) | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 2
Oedema peripheral (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 19 | 18 | 37
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 1
Acute graft versus host disease (Immune system disorders) | 1 | 1 | 2
Acute graft versus host disease in skin (Immune system disorders) | 0 | 1 | 1
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 1
Allergy to immunoglobulin therapy (Immune system disorders) | 0 | 1 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 1 | 2
Aspergillus infection (Infections and infestations) | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 1
Blastocystis infection (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 4 | 3 | 7
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 5 | 6
Campylobacter colitis (Infections and infestations) | 0 | 1 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 5 | 7
Chronic sinusitis (Infections and infestations) | 2 | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 1 | 1 | 2
Cytomegalovirus viraemia (Infections and infestations) | 0 | 2 | 2
Device related infection (Infections and infestations) | 1 | 0 | 1
Device related sepsis (Infections and infestations) | 2 | 0 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 1
Endocarditis (Infections and infestations) | 0 | 1 | 1
Endocarditis enterococcal (Infections and infestations) | 0 | 1 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 1 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 1 | 2
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1 | 1
Epididymitis (Infections and infestations) | 0 | 1 | 1
Epiglottitis (Infections and infestations) | 0 | 1 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 2
Gastrointestinal fungal infection (Infections and infestations) | 0 | 1 | 1
Genital herpes (Infections and infestations) | 0 | 1 | 1
H1N1 influenza (Infections and infestations) | 1 | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 3 | 4 | 7
Herpes zoster disseminated (Infections and infestations) | 1 | 0 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 4 | 1 | 5
Intervertebral discitis (Infections and infestations) | 1 | 2 | 3
JC virus infection (Infections and infestations) | 0 | 1 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 1
Leishmaniasis (Infections and infestations) | 0 | 1 | 1
Listeria sepsis (Infections and infestations) | 0 | 1 | 1
Listeriosis (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Lung infection (Infections and infestations) | 5 | 3 | 8
Meningitis (Infections and infestations) | 0 | 1 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1 | 1
Meningitis pneumococcal (Infections and infestations) | 1 | 1 | 2
Mucormycosis (Infections and infestations) | 1 | 0 | 1
Mycobacterial infection (Infections and infestations) | 1 | 0 | 1
Neuroborreliosis (Infections and infestations) | 0 | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 1 | 2
Nocardiosis (Infections and infestations) | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1 | 1
Parvovirus infection (Infections and infestations) | 0 | 1 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 0 | 2
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 2 | 2
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 1 | 3
Pneumonia (Infections and infestations) | 37 | 35 | 72
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1 | 1
Post procedural infection (Infections and infestations) | 1 | 0 | 1
Post procedural pneumonia (Infections and infestations) | 1 | 0 | 1
Post procedural sepsis (Infections and infestations) | 1 | 0 | 1
Postoperative abscess (Infections and infestations) | 0 | 1 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 1
Pulmonary sepsis (Infections and infestations) | 2 | 0 | 2
Respiratory tract infection (Infections and infestations) | 4 | 4 | 8
Sepsis (Infections and infestations) | 8 | 5 | 13
Septic shock (Infections and infestations) | 5 | 3 | 8
Sinusitis (Infections and infestations) | 3 | 2 | 5
Skin infection (Infections and infestations) | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 1 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 6
Urinary tract infection (Infections and infestations) | 3 | 5 | 8
Varicella (Infections and infestations) | 1 | 1 | 2
Varicella zoster virus infection (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 3 | 6
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Arthroscopy (Investigations) | 1 | 0 | 1
Calcium ionised increased (Investigations) | 1 | 0 | 1
Capillary permeability increased (Investigations) | 1 | 0 | 1
Heart rate irregular (Investigations) | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0 | 2
International normalised ratio increased (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypermetabolism (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Extraskeletal myxoid chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 4
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 0 | 2
Paraparesis (Nervous system disorders) | 0 | 1 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Toxic neuropathy (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Device dislocation (Product Issues) | 1 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Psychomotor retardation (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 2 | 2
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 1 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 2
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Allogenic bone marrow transplantation therapy (Surgical and medical procedures) | 1 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 1 | 1
Mastectomy (Surgical and medical procedures) | 0 | 1 | 1
Nasal septal operation (Surgical and medical procedures) | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 3
Haematoma (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Peripheral artery aneurysm (Vascular disorders) | 2 | 1 | 3
Venoocclusive disease (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=239) | Observation (N=241) | Total (N=480)
Neutropenia (Blood and lymphatic system disorders) | 61 | 22 | 83
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 11 | 24
Constipation (Gastrointestinal disorders) | 13 | 11 | 24
Diarrhoea (Gastrointestinal disorders) | 41 | 13 | 54
Nausea (Gastrointestinal disorders) | 13 | 8 | 21
Fatigue (General disorders) | 33 | 22 | 55
Oedema peripheral (General disorders) | 12 | 10 | 22
Pyrexia (General disorders) | 41 | 23 | 64
Hypogammaglobulinaemia (Immune system disorders) | 12 | 2 | 14
Bronchitis (Infections and infestations) | 21 | 17 | 38
Herpes zoster (Infections and infestations) | 14 | 8 | 22
Influenza (Infections and infestations) | 16 | 10 | 26
Nasopharyngitis (Infections and infestations) | 22 | 22 | 44
Pneumonia (Infections and infestations) | 17 | 11 | 28
Respiratory tract infection (Infections and infestations) | 17 | 15 | 32
Rhinitis (Infections and infestations) | 14 | 4 | 18
Sinusitis (Infections and infestations) | 22 | 9 | 31
Upper respiratory tract infection (Infections and infestations) | 52 | 26 | 78
Infusion related reaction (Injury, poisoning and procedural complications) | 42 | 0 | 42
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 12 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 12 | 27
Headache (Nervous system disorders) | 23 | 7 | 30
Insomnia (Psychiatric disorders) | 14 | 6 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 28 | 86
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 9 | 32
Rash (Skin and subcutaneous tissue disorders) | 26 | 10 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT01039376/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT01039376/SAP_002.pdf